CLINICAL TRIAL: NCT01583400
Title: Development and Evaluation of Enhanced Digital Health Coaching Program for Depressive Symptoms to Support Collaborative Depression Treatment in Primary Care: The RESPECT-D-E (Enhanced) Trial
Brief Title: Enhanced Collaborative Depression Treatment in Primary Care: The RESPECT-D-E Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Mark T. Hegel, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPHS#22616, W&P-PCMH-01
Record Dates: First submitted 2012-04-12; First posted 2012-04-24 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Depressive Disorder, Major; Depressive Disorder, Minor; Dysthymic Disorder
Keywords: Depressive Disorder, Major; Depressive Disorder, Minor; Dysthymic Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Dysthymic Disorder | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RESPECT-D (Active Comparator): The RESPECT-D Model: Collaborative Care depression treatment within primary care including care manager
  Interventions: Other: RESPECT-D
- RESPECT-D-E (Experimental): RESPECT-D-E: Collaborative Care depression treatment within primary care including care manager plus on-line coaching, education and symptom, side effect and, medication adherence tracking with the digital health coaching program for depressive symptoms.
  Interventions: Other: RESPECT-D-E (Enhanced)

INTERVENTIONS:
Other: RESPECT-D — The RESPECT-D (Re-engineering Systems of Primary Care Treatment of Depression) intervention is a systematic approach to the assessment and management of depression within Primary Care. The essential components of the Collaborative Care model include prepared PCPs and practices, the Care Manager, and a Behavioral Health specialist all working in partnership with the patient. The trained depression care manager closely coordinates with primary care clinicians, supports treatment recommendations, patient education, appropriate follow-up to ensure adequate treatment, and coordination with a consulting psychiatrist.
  Other Names: Collaborative Care Treatment for Depression in Primary Care
  Arms: RESPECT-D
Other: RESPECT-D-E (Enhanced) — The RESPECT-D-E intervention includes all of the components of the RESPECT-D model, but also incorporates the enhanced digital health coaching program for depressive symptoms tool, is an on-line program with education, coaching, self-management techniques, symptom, side effect and medication adherence tracking for depression. Depressive symptoms, medication side effects and adherence data are automatically delivered to the Care Manager for use in treatment planning. The program provides tailored feedback, provides coaching on skills related to depression treatment (such as changing negative thoughts and avoiding relapse), and offers tools for tracking behavior change.
  Other Names: Enhanced Collaborative Care Treatment for Depression in Primary Care; Digital Health Coaching Program for Depressive Symptoms
  Arms: RESPECT-D-E

SUMMARY:
Primary care physicians have emerged as the predominant mental health care providers for diagnosing and treating depression. The majority of patients with mood disorders receive treatment in the primary care setting, within which approximately 10-30% of all patients present with a depressive disorder. Comprehensive 'Collaborative Care' models of depression management significantly improve depression outcomes and health-related quality of life. Core features of these programs include use of a trained depression care manager to closely coordinate with primary care clinicians, support treatment recommendations, provide patient education, conduct patient follow-up to ensure adequate treatment, and manage as-needed access to psychiatrists for patients with more complex presentations. Evidence based Collaborative Care models do not currently weave in the use of web-based or mobile technologies. These technologies offer unique features that may make collaborative depression care more effective. The digital health coaching program for depressive symptoms enhanced during Phase I of the current project is a web-based tool featuring video, text, links and graphics which provide patients with education, self-management techniques, tailored feedback, and tools for tracking treatment progress. The RESPECT-D (Re-engineering Systems of Primary Care Treatment of Depression) intervention is a collaborative depression management model for primary care. The primary objective of this project is to compare the efficacy of an enhanced Collaborative Care model for depression (RESPECT-D-E) to the standard model (RESPECT-D) for patients with minor and major depression and dysthymic disorder. This study will be a randomized controlled trial with 150 participants who are receiving antidepressant medication treatment in the primary care setting. The primary objectives are: reduction in subject reported depressive symptoms, improvement in subject reported health related quality of life and improvement in subject adherence to treatment regimen as demonstrated by self-report measures and clinician-administered assessment. The investigators hypothesize that compared to RESPECT-D at 12 weeks, participants randomized to RESPECT-D-E will demonstrate: a greater reduction in depressive symptoms, a greater improvement in health-related quality of life and a greater satisfaction with quality of depression care received.

DETAILED DESCRIPTION:
The National Comorbidity Survey suggests a lifetime prevalence of 17% and 1-year prevalence of 10% for major depression. Within primary care, approximately 10-30% of patients present with a depressive disorder. Over the past decade, primary care physicians have emerged as the predominant mental health care providers insofar as diagnosing and treating depression, with the majority of patients with mood disorders receiving treatment in a primary care setting.

Comprehensive 'Collaborative Care' models of depression management in primary care significantly improve depression outcomes and health-related quality of life. Core features of these programs include use of a trained depression care manager to closely coordinate with primary care clinicians, provision of specific treatment recommendations/guidelines, patient education, appropriate follow-up by the depression care manager to ensure adequate treatment, as-needed access to psychiatrists for patients with more complex presentations, and, occasionally, on-site psychotherapy. For example, the IMPACT study of primary care patients with late-life depression found that a Collaborative Care program doubled the effectiveness of depression treatment and improved functional outcomes at 3 months, 6 months and 1 year compared to usual care. The RESPECT-D phone-based Collaborative Care program similarly had increases at 3 and 6 months in depression response, remission, and satisfaction with care, compared to usual care.

Nonetheless, evidence based Collaborative Care leaves room for improvement. In both IMPACT and RESPECT-D, 40% to 50% of intervention participants failed to achieve a clinically meaningful depression treatment effect. Evidence based Collaborative Care models do not currently weave in the use of web-based or mobile technologies. These technologies offer unique features that may make collaborative depression care more effective. The enhanced digital health coaching program for depressive symptoms is a web-based tool featuring video, text and graphics which provides patients with education, self-management techniques, tailored feedback, and tools for tracking treatment progress. Incorporating a digital health coaching program for depressive symptoms into the flow of collaborative depression care and testing its impact is an important next step for the field.

The RESPECT-D (Re-engineering Systems of Primary Care Treatment of Depression) intervention is a systematic approach to the assessment and management of depression by the primary care provider, with a centrally based care manager providing telephone support for patients. The essential components of this Collaborative Care model include prepared PCPs and practices, the Care Manager, and a Behavioral Health specialist all working in partnership with the patient.

RESPECT-D-E (Enhanced) intervention is Collaborative Care depression treatment in primary care including care manager (the elements of RESPECT-D) plus patient access to on-line coaching, education, and symptom, side effect and medication adherence tracking which is automatically fed back to the Care Manager.

The primary objective of this project is to compare the efficacy of an enhanced Collaborative Care model for depression (RESPECT-D-E) to the standard model (RESPECT-D) in primary care patients with minor and major depression and dysthymic disorder .

The RESEPCT-D-E trial is a randomized, 12-week prospective 2-arm, comparative clinical effectiveness study. Primary care patients (N=150) with major or minor depressive disorder, or dysthymia and currently taking antidepressant medication will be randomly assigned to either Collaborative Care treatment for depression (RESPECT-D) or RESPECT-D plus a digital health coaching program for depressive symptoms intervention (RESPECT-D-E). Patients will be assessed at baseline, 4 weeks, 8 weeks, and 12 weeks using self-report and clinician -administered rating scales including the Hopkins Symptom Checklist and Hamilton Depression Rating Scale. Intervention participants will receive access to the online depression coach as well as the elements of standard Collaborative Care (RESPECT-D). The primary objectives are: reduction in depressive symptoms, improvement in health related quality of life and improvement in adherence to treatment regimen.

The secondary objectives of the RESPECT-D-E trial are to: Evaluate the program impact on overall health, work productivity, and medical costs; Assess the usability of the enhanced digital health coaching program for depressive symptoms tool; Assess the program's impact on overall satisfaction with care.

Hypotheses: Compared to RESPECT-D at 12 weeks, participants randomized to RESPECT-D-E will demonstrate: H1.1a: a greater reduction in depressive symptoms, as measured by the clinician administered Hamilton Depression Rating Scale (HAM-D); H1.1b: a greater reduction in depressive symptoms, as measured by the self-report Hopkins Symptom Checklist Depression Scale (HSCL-20); H1.1c: a greater improvement in health related quality of life, as measured by the Mental Component Summary score from the Medical Outcomes Study Short Form (SF-36); H1.1d: a greater satisfaction with quality of depression care received.

Hypothesis 1.2: Compared to RESPECT-D at 4, 8, and 12 weeks, participants randomized to RESPECT-D-E will demonstrate: H1.2a: more frequent contact with the depression care manager and primary care provider, as measured by depression care manager treatment logs and medical record review; H1.2b: greater adherence to their antidepressant regimen, as measured by participant self-report; H1.2c: greater exposure to depression counseling, as measured by participant self-report.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, ages 18 and older who are self-reporting generally good health.
* Newly started on an antidepressant medication, switched to a different antidepressant medication or prescribed an increased dosage of antidepressant medication within the past 2 weeks.
* A Hamilton Depression Rating Scale (HAM-D) score of greater than 10.
* A Patient Health Questionnaire (PHQ-9) score of 10 or greater, with endorsement of depressed mood or anhedonia, and endorsement of impaired daily function.
* Meets diagnostic criteria for Major Depressive Disorder, persistent Minor Depressive Disorder (i.e., > 1 month duration), or Dysthymic Disorder via a structured interview with the PRIME-MD.
* Able to read, understand, and sign the Informed Consent in English.
* Willing and able to comply with study requirements.
* Well-versed in using a personal computer and the internet and must have easy access to a computer connected to the internet everyday (both weekdays and weekends).
* Enrollment in Surescripts Pharmacy benefit plan
* Currently under care with a Provider in Family Medicine at Cheshire Medical Center / Dartmouth-Hitchcock Keene

Exclusion Criteria:

* Subjects must not have a major psychiatric co-morbid condition (schizophrenia, bipolar affective disorder, obsessive-compulsive disorder, PTSD, or a depressive disorder with psychotic features, as determined from chart review and patient report).
* Subjects must not have a substance use disorder or dependence as assessed by: CAGE Alcohol Dependence Questionnaire score >3
* Subjects must not have a history of treatment -resistant depression as defined by the following: Psychiatric hospitalization within the past year; More than 2 clinically ineffective antidepressant medication trials, of adequate duration and adequate dose, within the current depressive episode; Any history of Electroconvulsive Therapy (ECT); A trial of Monoamine Oxidase inhibitor (MAO) within the past year.
* Subjects must not report being actively suicidal
* Subjects must score 4 or greater on the Callahan Six-Item Cognitive Screening assessment
* Subjects must not be diagnosed with a terminal or near terminal medical illness such that their primary care provider has estimated the patient has less than 6 months to live.
* Subjects reporting any medical condition that would make it unsafe to participate in a research study.
* Participation in any other clinical research study within the past 30 days.
* Participation in any on-line depression-related coaching or lifestyle improvement program within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Score of Hamilton Rating Scale for Depression (HAM-D) | 12 weeks
  17-item assessment rated during a clinical interview

SECONDARY OUTCOMES:
Change in Score of Hopkins Symptom Checklist-20 (HSCL-20) | 12 weeks
  Self-report measure of depressive symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Mark T. Hegel, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Family Medicine Clinics, Cheshire Medical Center (DH-Keene), Keene, New Hampshire, United States

REFERENCES:
- [Background] Dietrich AJ, Oxman TE, Williams JW Jr, Schulberg HC, Bruce ML, Lee PW, Barry S, Raue PJ, Lefever JJ, Heo M, Rost K, Kroenke K, Gerrity M, Nutting PA. Re-engineering systems for the treatment of depression in primary care: cluster randomised controlled trial. BMJ. 2004 Sep 11;329(7466):602. doi: 10.1136/bmj.38219.481250.55. Epub 2004 Sep 2. PMID 15345600
- [Background] Hunkeler EM, Katon W, Tang L, Williams JW Jr, Kroenke K, Lin EH, Harpole LH, Arean P, Levine S, Grypma LM, Hargreaves WA, Unutzer J. Long term outcomes from the IMPACT randomised trial for depressed elderly patients in primary care. BMJ. 2006 Feb 4;332(7536):259-63. doi: 10.1136/bmj.38683.710255.BE. Epub 2006 Jan 20. PMID 16428253
- [Background] Katon W, Von Korff M, Lin E, Walker E, Simon GE, Bush T, Robinson P, Russo J. Collaborative management to achieve treatment guidelines. Impact on depression in primary care. JAMA. 1995 Apr 5;273(13):1026-31. PMID 7897786
- [Background] Katon WJ, Von Korff M, Lin EH, Simon G, Ludman E, Russo J, Ciechanowski P, Walker E, Bush T. The Pathways Study: a randomized trial of collaborative care in patients with diabetes and depression. Arch Gen Psychiatry. 2004 Oct;61(10):1042-9. doi: 10.1001/archpsyc.61.10.1042. PMID 15466678
- [Background] Katon W, Von Korff M, Lin E, Simon G, Walker E, Unutzer J, Bush T, Russo J, Ludman E. Stepped collaborative care for primary care patients with persistent symptoms of depression: a randomized trial. Arch Gen Psychiatry. 1999 Dec;56(12):1109-15. doi: 10.1001/archpsyc.56.12.1109. PMID 10591288
- [Background] Torrey WC, Drake RE. Practicing shared decision making in the outpatient psychiatric care of adults with severe mental illnesses: redesigning care for the future. Community Ment Health J. 2010 Oct;46(5):433-40. doi: 10.1007/s10597-009-9265-9. Epub 2009 Nov 8. PMID 19898985
- [Background] Unutzer J, Katon W, Callahan CM, Williams JW Jr, Hunkeler E, Harpole L, Hoffing M, Della Penna RD, Noel PH, Lin EH, Arean PA, Hegel MT, Tang L, Belin TR, Oishi S, Langston C; IMPACT Investigators. Improving Mood-Promoting Access to Collaborative Treatment. Collaborative care management of late-life depression in the primary care setting: a randomized controlled trial. JAMA. 2002 Dec 11;288(22):2836-45. doi: 10.1001/jama.288.22.2836. PMID 12472325
- [Background] Kessler RC, Nelson CB, McGonagle KA, Liu J, Swartz M, Blazer DG. Comorbidity of DSM-III-R major depressive disorder in the general population: results from the US National Comorbidity Survey. Br J Psychiatry Suppl. 1996 Jun;(30):17-30. PMID 8864145
- [Background] McQuaid JR, Stein MB, Laffaye C, McCahill ME. Depression in a primary care clinic: the prevalence and impact of an unrecognized disorder. J Affect Disord. 1999 Sep;55(1):1-10. doi: 10.1016/s0165-0327(98)00191-8. PMID 10512600
- [Background] Norquist GS, Regier DA. The epidemiology of psychiatric disorders and the de facto mental health care system. Annu Rev Med. 1996;47:473-9. doi: 10.1146/annurev.med.47.1.473. PMID 8712797
- [Background] Stein MB, Kirk P, Prabhu V, Grott M, Terepa M. Mixed anxiety-depression in a primary-care clinic. J Affect Disord. 1995 May 17;34(2):79-84. doi: 10.1016/0165-0327(95)00002-5. PMID 7665808
- [Background] Weilburg JB, O'Leary KM, Meigs JB, Hennen J, Stafford RS. Evaluation of the adequacy of outpatient antidepressant treatment. Psychiatr Serv. 2003 Sep;54(9):1233-9. doi: 10.1176/appi.ps.54.9.1233. PMID 12954939